CLINICAL TRIAL: NCT06286943
Title: The Effects of Gut Bacterial Metabolites Short-Chain Fatty Acids on Stress-Induced Impairment in Core Executive Functions
Brief Title: The Effects of Short-Chain Fatty Acids in Psychosocial Stress-Induced Impairment on Core Executive Functions
Acronym: GUTSIE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: S68124
Record Dates: First submitted 2024-02-16; First posted 2024-02-29 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-02

CONDITIONS: Executive Function
MeSH Terms: interventions — Fatty Acids, Volatile; Cold Temperature

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Microcrystalline cellulose placebo capsules.
  Interventions: Dietary Supplement: Placebo; Other: Maastricht Acute Stress Task; Other: No-stress control task
- SCFAs (Experimental): Colon-delivery Capsules of Short Chain Fatty Acids.
  Interventions: Dietary Supplement: Short Chain Fatty Acids (SCFAs).; Other: Maastricht Acute Stress Task; Other: No-stress control task

INTERVENTIONS:
Dietary Supplement: Short Chain Fatty Acids (SCFAs). — Colon-delivery capsules of SCFAs.
  Arms: SCFAs
Dietary Supplement: Placebo — Microcrystaline cellulose placebo capsules.
  Arms: Placebo
Other: Maastricht Acute Stress Task — The Maastricht Acute Stress Task. This 15-minute stress-inducing task consists of a 5-minute preparation phase where instructions about the upcoming tasks are given, followed by a 10-minute acute stress phase where the hand immersion trial (HIT) in ice-cold water and mental arithmetic (MA) task is given interchangeably.
  Other Names: MAST, cold, arithmetics
Other: No-stress control task — The placebo version of the MAST follows the same structure of the MAST with none of the stress elements. It uses lukewarm water and simple arithmetic's.
  Other Names: Sham MAST

SUMMARY:
The aim of the present trial is to examine core executive functions (EFs) as a functional outcome of attenuating the cortisol response to acute laboratory stress through colonic delivery of an Short Chain Fatty Acids (SCFAs) mix (acetate, propionate, butyrate).

A triple-blind randomized placebo-controlled parallel group trial will be conducted to compare the effects of SCFAs vs. placebo on core EFs (working memory [WM], cognitive flexibility [CF], response inhibition [RI]) under stress vs. no-stress conditions, after one week of SCFA vs. placebo treatment.

First, the effects of SCFAs on stress-induced changes in core executive functions, with WM as the primary outcome, and CF and RI as secondary outcomes will be tested. Second, interindividual differences in microbiota composition (particularly abundance of SCFA-producers), saliva cortisol and serum SCFA levels will be explored to assess whether they are associated with interindividual differences in core EFs at baseline or following acute stress.

Each participant will undergo 2 study visits: one will involve a stress condition and the other will involve a no-stress condition. Each study visit is preceded by a 1-week intervention or placebo period and separated by a 3-4 week washout period. To induce stress, participants will perform the Maastricht Acute Stress Task (MAST) or sham MAST as the control condition. To assess EF performance, three cognitive tasks will be performed 15 minutes after task offset: n-back task for WM; Stop Signal Task for RI; and Wisconsin Card Sorting Test for CF. Saliva samples will be collected before, during and after the (sham) MAST to assess the cortisol response. Blood samples will be collected throughout all study visits to quantify serum SCFAs, inflammatory markers and ACTH. Additionally, cardiovascular variables will be measured, and self-report questionnaires will be completed to evaluate autonomic response to the condition and subjective stress responses, respectively

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
* Proficiency in English and/or Dutch
* Healthy with no intestinal and/or psychological complaints
* Access to a -18°C freezer (i.e. ordinary household freezer)
* Male participants
* Age 20-40 years
* BMI 18.5-25 kg/m2

Exclusion Criteria:

* Participant has a history of previous or current neurological, psychiatric, gastrointestinal or endocrine disorder
* Any disorder, which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol
* Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the study
* Participation in an interventional Trial with an investigational medicinal product (IMP) or device
* Current or recent (over the past month) medication use as a (prescribed) medical treatment. This does not include isolated intakes of 'over the counter' medication (e.g. ibuprofen, paracetamol).
* Use of antibiotics within three months preceding the study.
* Current or recent (1-month) infection (e.g. common cold, influenza, COVID-19, etc.)
* Recent (1-month) vaccination (e.g. flu shot, SARS-COV-2 vaccine, etc)
* Previous or current substance/alcohol dependence or abuse (>2 units per day or 14 units per week).
* One or more diagnoses based on the Mini International Neuropsychiatric Interview.
* One or more diagnoses based on ROME-IV for gastrointestinal disorders.
* Smoking.
* Night-shift work.
* Adherence to special diets (e.g. vegan, vegetarian, weight-loss, lactose-free, gluten-free, etc.).
* Use of pre- or probiotics within one month preceding the study.
* Previous experience with or knowledge of any of the tasks used in the study (not including questionnaires).

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Working memory | Test day 1 and Test day 2 (Stress vs. No-stress conditions)
  n-Back task

SECONDARY OUTCOMES:
Cognitive Flexibility | Test day 1 and Test day 2 (Stress vs. No-stress conditions)
  Wisconsin Card Sorting Task
Response Inhibition | Test day 1 and Test day 2 (Stress vs. No-stress conditions)
  Stop Signal Task